CLINICAL TRIAL: NCT00116285
Title: A Single-Blind Phase I Study to Assess the Residual Allergenicity of Tyrosine Adsorbed Ragweed Pollen Allergoid With MPL Using Skin Prick Testing
Brief Title: Assessment of Residual Allergenicity of Ragweed Pollen Allergoid With Monophosphoryl Lipid A (MPL) Using Skin Prick Testing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RagweedMATAMPL101; P1DP05003
Record Dates: First submitted 2005-06-28; First posted 2005-06-29 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2009-09

CONDITIONS: Type I Hypersensitivity
Keywords: allergy; skin prick test; allergoid; allergenicity; specific immunotherapy
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity | interventions — ragweed MATA MPL

INTERVENTIONS:
Biological: Ragweed MATA MPL

SUMMARY:
The purpose of this study is to evaluate the residual allergenicity of the modified ragweed pollen in Ragweed MATA MPL (modified pollen allergen tyrosine adsorbate + Monophosphoryl Lipid A) by skin prick testing. This is done by a comparison of the wheal response after skin prick testing with different concentrations of aqueous native allergen, modified allergen, modified tyrosine adsorbed allergen, and Ragweed MATA MPL.

DETAILED DESCRIPTION:
Ragweed MATA MPL has been developed to provide pre-seasonal specific immunotherapy for patients with proven type I hypersensitivity to ragweed pollen. MPL (Monophosphoryl Lipid A), a purified, detoxified glycolipid derived from the cell wall of Salmonella minnesota, is included in the product formulation as an adjuvant to increase the immunogenic effect of the product and to enhance the switch from an allergen-specific TH2 to a TH1-like profile.

The ragweed pollen extract is modified with glutaraldehyde to produce the active ingredient, an allergoid. This modification reduces the reactivity of the extract with IgE antibody, thus reducing the risk of side effects. However, a simultaneous reduction in other important immunological properties, such as IgG and T cell reactivities is not seen.

The purpose of this study is to assess residual allergenicity of the modified ragweed pollen in Ragweed MATA MPL using skin prick testing.

ELIGIBILITY:
Inclusion Criteria:

* If the volunteer is female of childbearing potential, she must demonstrate a negative urine pregnancy test and agree to remain abstinent or use an effective method of birth control
* Positive skin prick test to ragweed pollen allergen extract
* Positive skin prick test to positive histamine control
* Negative skin prick test to negative control; redness, but no wheal is acceptable
* The subject must demonstrate a specific IgE for ragweed with class >= 2.
* The subject must have clinically acceptable results from the screening procedure including blood pressure (BP), heart rate (HR), electrocardiogram (ECG), physical examination, medical history, hematology, biochemistry, infection screen (hepatitis B antigen, hepatitis C antibody, HIV), urine pregnancy test, urinalysis, drugs of abuse screening panel and saliva alcohol testing

Exclusion Criteria:

* History or presence of acute or subacute atopic dermatitis, chronic dermatitis, urticaria factitia, or urticaria due to physical/chemical influence or any other skin conditions which might interfere with the interpretation of skin prick test results
* Visual inspection of the forearms indicates potential problems with the conduct or interpretation of the skin prick tests; both forearms must be available for testing
* Subject has asthma or other lower respiratory tract condition
* History or presence of diabetes, cancer or any clinically significant cardiac, metabolic, renal, hepatic, gastrointestinal, dermatologic, venereal, hematologic, neurologic or psychiatric diseases or disorders
* Any clinically significant abnormal laboratory value at Visit 1
* Clinically relevant sensitivity to any of the following common perennial or seasonal allergens: house dust mites, molds, epithelia, grass pollen mix, plantain, orache, nettle, mugwort, bermuda grass
* Clinically relevant symptoms due to an IgE-mediated allergy at screening and before inclusion to the treatment period
* Secondary alteration at the affected organ
* History of auto-immune diseases or rheumatoid diseases
* Medical condition that prohibits the use of adrenaline
* Disorder of tyrosine metabolism
* Diseases interfering with the immune response and having received medication which could influence the results of this study
* Subject has acute or chronic infection
* History of anaphylaxis
* Subjects determined by the Investigator to have any medical condition that could jeopardize their health or prejudice the results
* History of hypersensitivity to the excipients of the study medication
* History of immunotherapy with ragweed allergen extracts
* Current therapy with ß-blockers
* Currently receiving anti-allergy medication or other drugs with an antihistaminic activity
* Subject has a positive drugs of abuse screen at Visit 1
* Subject participated in a clinical trial and has taken investigational drug within the last 30 days
* Subject cannot communicate reliably with the Investigator or is deemed uncooperative or noncompliant
* Females who are pregnant, breastfeeding, or refuse to use a reliable method of birth control
* Subject received treatment with a preparation containing MPL during the past 12 months
* Use of prohibited medications or inadequate washout periods prior to screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12
Dates: Start 2005-06; Study Completion 2005-06

PRIMARY OUTCOMES:
To assess the allergenicity of the modified ragweed pollen in Ragweed MATA MPL compared to unmodified native allergen using skin prick testing

SECONDARY OUTCOMES:
To assess the safety and tolerability of the skin prick test products

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, Principal Investigator — Allied Research International Inc.
Locations (1):
- Allied Research International Inc., Mississauga, Ontario, Canada